CLINICAL TRIAL: NCT06457789
Title: Assessment of PET Tracers to Evaluate T Cell Change and Activation in Relation to Immunotherapy Treatment Response in Non-Small Cell Lung Cancer
Acronym: iRelate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Foundation for the National Institutes of Health (Other)
Responsible Party: Principal Investigator, Idris Bahce, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-509486-20-00; 2023-509486-20-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-03; First posted 2024-06-13 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: NSCLC
Keywords: NSCLC; immunoPET; 18F-AraG; AraG; 89Zr-crefmirlimab; Crefmirlimab; tracers; PET tracers; [18F]F-AraG; [89Zr]Zr-Df-Crefmirlimab; IAB22M2C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual T cell PET imaging (Experimental): Patients will receive PET imaging with two different T-cell targeting tracers.
  Interventions: Drug: [18F]F-AraG PET imaging; Drug: [89Zr]Zr-Df-Crefmirlimab PET imaging

INTERVENTIONS:
Drug: [18F]F-AraG PET imaging — Patients will receive a static whole-body PET scan following a [18F]F-AraG injection.
Drug: [89Zr]Zr-Df-Crefmirlimab PET imaging — Patients will receive a static whole-body PET scan following a [89Zr]Zr-Df-Crefmirlimab injection.

SUMMARY:
The iRelate is a PET imaging trial to compare two upcoming and promising T cell PET tracers. Following chemo-immuno therapy, as part of standard care, NSCLC patients will be recruited to receive two PET scans, shortly before their surgery. Both PET scans will be compared to each other, as well as compared to the pathological analysis of the resected tumor.

This study will provide detailed information on the unique as well as additive capacities of imaging biomarkers derived from the immune cell targeting PET tracers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC
* T1-4N0-2, lesion size of ≥2cm, at time of the restaging FDG PET/CT
* Planned to undergo resection after chemo-IO according to routine treatment guidelines
* Willing and able to provide written informed consent for the trial
* Above 18 years of age on day of signing informed consent
* Have measurable disease based on RECIST 1.1
* Have a ECOG performance status of 0-1, and are considered operable based on pulmonary function test and/or exercise testing

Exclusion Criteria:

* Patients deemed inoperable
* Patients who have received a splenectomy
* Patients who have received any vaccination within 14 days of enrollment
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of day 0. Inhaled or topical steroids, and adrenal replacement steroid >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patient is pregnant or breastfeeding or expecting to conceive within the projected duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
To measure the spatial correlation of PET uptake of [18F]F-AraG and [89Zr]Zr-Df-Crefmirlimab in tumors and T-cell rich organs such as lymph nodes prior to resection. | 2 months
  The spatial overlap of the regions of uptake for both PET tracers will be assessed using the Dice Similarity Coefficient (DSC) as an established method
To measure the strength of correlation between the presence of CD8+ cells and T cell activation features in the resected tumor and lymph nodes with preoperative uptake of [89Zr]Zr-Df-Crefmirlimab and [18F]F-AraG, respectively. | 6 months
  The Pearson correlation coefficient between each tracer tumor uptake and the T cell features in regions of concordance and discordance.

SECONDARY OUTCOMES:
To measure the strength of correlation of pathological response (i.e., the residual viable tumor cells percentage) in the resected tumor with preoperative uptake of [89Zr]Zr-Df-Crefmirlimab and [18F]F-AraG. | 6 months
  The Pearson correlation coefficient between each tracer tumor uptake and percentage of residual viable tumor cells (VTC) in regions of concordance and discordance and the maximal VTC of the entire tumor. The Pearson correlation coefficient between each tracer uptake and the T cell presence in resected lymph nodes (if present).

OTHER OUTCOMES:
To explore the association of PET uptake of both tracers in tumor and T-cell rich organs such as lymph nodes with: The immune profile of the TME and resected lymph nodes beyond T cells. The immune profile of peripheral blood mononuclear cells (PBMCs) | 6 months
  The Pearson correlation coefficient between PET uptake and immune profile of the TME for tumor and T-cell rich organs. The Pearson correlation coefficient between PET uptake and immune profile of PBMCs for tumor + T-cell rich organs.
To quantify inter- and intra-tumoral heterogeneity of PET tracer uptake. | 2 months
  Voxel intensities for [18F]F-AraG and [89Zr]Zr-Df-Crefmirlimab PET images will be plotted against each other by means of scatter plots and joint histograms/kernel density plots to illustrate the degree of agreement in spatial distribution of both tracers with the VOIs.
To assess the relationship of metabolically active areas as assessed by [18F]F-FDG PET with areas of uptake derived from [18F]F-AraG and [89Zr]Zr-Df-Crefmirlimab PET. | 4 months
  The spatial overlap of the regions of uptake for the FDG, [18F]F-AraG and [89Zr]Zr-Df-Crefmirlimab PET tracers will be assessed using the Dice Similarity Coefficient (DSC) method.

CONTACTS AND LOCATIONS:
Overall Officials: Idris Bahce, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided